CLINICAL TRIAL: NCT03717727
Title: Effectiveness of Gamification in Knee Replacement Rehabilitation. Randomized Controlled Trial and Qualitative Approach
Brief Title: Gamification in Knee Replacement Rehabilitation
Acronym: BEE-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Turku University Hospital (Other Government); Turku University of Applied Sciences (Unknown); Jyväskylä Central Hospital (Other); University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T226/2018
Record Dates: First submitted 2018-10-08; First posted 2018-10-24 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee replacement; Exergame; Total knee arthroplasty; Exercise; Physiotherapy; Physical functioning
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame (Experimental): Home-based exergame intervention and usual treatment.
  Interventions: Other: Exergame
- Control (Experimental): Home-exercise by standard protocol and usual treatment.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exergame — 16-week home-based exercise intervention with exergaming system and usual treatment.
  Other Names: Gamified rehabilitation
  Arms: Exergame
Other: Control — 16-week home-based exercise by standard protocol and usual treatment.
  Arms: Control

SUMMARY:
After total knee arthroplasty (TKA), knee is usually swollen, painful, and stiff. The main goal of post-operative physical rehabilitation is to achieve full extension and flexion of the knee to avoid contractures and stiffness. Also strengthening of quadriceps muscle and balance to help activities of daily living and overall mobility are important. The post-operative knee replacement rehabilitation includes the standard protocol in hospital phase and the standard home exercise instructions. Computer based exercising games (exergames) may be new method to increase training adherence and volume after TKA and thus improve results and effectiveness of the rehabilitation. However, evidence of effectiveness of rehabilitative exergaming on physical functioning is sparse and more research is needed to conduct evidence-based rehabilitation practices.

Therefore the present study examines the effectiveness of a 16-week gamified physiotherapy on physical functioning, life satisfaction and pain for patients after TKA compared to treatment as usual home exercise. The second objective is to validate the psychometric properties of WHODAS 2.0 (WHO Disability Assessment Schedule) and brief ICF (International classification of functioning, disability and health) core set of osteoarthritis questionnaire. Other objectives are to find out, what kind of understanding and experiences the participants have about the rehabilitation with exergames and to evaluate the usability and user experience of exergames.

ELIGIBILITY:
Inclusion Criteria:

* first primary (M17.0, M17.1) unilateral TKA
* mechanical axis of the limb in varus
* model of the TKA is posterior stabilizing (PS) or cruciate retaining (CR) prosthesis
* normal vision with or without eyeglasses

Exclusion Criteria:

* fractures, rheumatoid arthritis, or other biomechanical disruptions in affected lower limb within one year before operation
* diagnosed memory disorder or cognitive impairment
* neurological condition as Parkinson's disease, multiple sclerosis or stroke

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Function and pain related to knee | Change from pre-operative baseline at 2 and 4 months post-operative.
  Oxford Knee Score
Change in Mobility | Change from pre-operative baseline at 2 and 4 months post-operative.
  Timed Up and Go

SECONDARY OUTCOMES:
Change in Function and pain related to knee | Change from pre-operative baseline at 12 months post-operative.
  Oxford knee score
Change in Mobility | Change from pre-operative baseline at 12 months post-operative.
  Timed Up and Go
Change in Walking | pre-operative baseline and 2, 4 and 12 months post-operative
  10-m Walking speed
Change in Lower extremity performance | pre-operative baseline and 2, 4 and 12 months post-operative
  Short Physical Performance Battery
Change in Muscle strength | pre-operative baseline and 2, 4 and 12 months post-operative
  Isometric knee extension and flexion strength
Change in Knee range of motion | pre-operative baseline and 2, 4 and 12 months post-operative
  Goniometer
Change in knee pain (VAS) | pre-operative baseline and 2, 4 and 12 months post-operative
  Visual analogue scale (0 to 100 mm), Constant score (0 to 100 points)
Change in Disability | pre-operative baseline and 2, 4 and 12 months post-operative
  WHO disability scale (WHODAS 2.0.)
Change in Pain | pre-operative baseline and 2, 4 and 12 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale on pain.
Change in other symptoms such as swelling, restricted range of motion and mechanical symptoms | pre-operative baseline and 2, 4 and 12 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale on symptoms
Change in quality of life (QOL) | pre-operative baseline and 2, 4 and 12 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale on QOL
Change in activities of daily living (ADL) Function | pre-operative baseline and 2, 4 and 12 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale on ADL
Change in Sport and Recreation Function | pre-operative baseline and 2, 4 and 12 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) subscale on Sport and Recreation Function

OTHER OUTCOMES:
Physical activity | Through study completion, an average of 1 year
  Physical activity diary
Satisfaction with the operated knee | 2, 4 and 12 months post-operative
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Keijo Mäkelä, Principal Investigator — Turku University Hospital; Ari Heinonen, Principal Investigator — University of Jyvaskyla
Locations (4):
- Finland (4):
  - Central Finland Central Hospital, Jyväskylä
  - University of Jyväskylä, Jyväskylä
  - Turku University Hospital, Turku
  - Turku University of Applied Sciences, Turku

IPD SHARING:
Plan to Share IPD: No
Sensitive parts of the data cannot be anonymized and thus cannot be openly published. Sensitive data will be stored in JYX (Jyväskylä University Digital Repository), only the metadata will be public, and access to the data can be requested and granted on certain conditions. Metadata published in the Jyväskylä University Digital Repository. Heinonen A, Janhunen M, Aarto-lahti E, et al. Metadata from: Gamification in Knee Replacement Rehabilitation (BEE-RCT). V.2.2.2023 doi:10.17011/jyx/dataset/85350

REFERENCES:
- [Background] Aartolahti E, Janhunen M, Katajapuu N, Paloneva J, Pamilo K, Oksanen A, Keemu H, Karvonen M, Luimula M, Korpelainen R, Jamsa T, Makela K, Heinonen A. Effectiveness of Gamification in Knee Replacement Rehabilitation: Protocol for a Randomized Controlled Trial With a Qualitative Approach. JMIR Res Protoc. 2022 Nov 28;11(11):e38434. doi: 10.2196/38434. PMID 36441574
- [Result] Janhunen M, Katajapuu N, Paloneva J, Pamilo K, Oksanen A, Keemu H, Karvonen M, Luimula M, Korpelainen R, Jamsa T, Kautiainen H, Makela K, Heinonen A, Aartolahti E. Effects of a home-based, exergaming intervention on physical function and pain after total knee replacement in older adults: a randomised controlled trial. BMJ Open Sport Exerc Med. 2023 Mar 3;9(1):e001416. doi: 10.1136/bmjsem-2022-001416. eCollection 2023. PMID 36896366
- See also: Primary results — https://bmjopensem.bmj.com/content/9/1/e001416
- See also: Study protocol — https://www.researchprotocols.org/2022/11/e38434/
- Available data/document: Metadata — https://doi.org/10.17011/jyx/dataset/85350 — Metadata published in the Jyväskylä University Digital Repository. Heinonen A, Janhunen M, Aartolahti E, et al. Metadata from: Gamification in Knee Replacement Rehabilitation (BEE-RCT)